CLINICAL TRIAL: NCT00879372
Title: Double Blind,Randomized, Placebo Controlled Trial of Adjunctive Tianeptine in the Treatment of Bipolar Depression
Brief Title: Efficacy of Adjunctive Tianeptine in the Treatment of Bipolar Depression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Flavio Kapczinski, PhD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-145
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; cognitive impairment; depression
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction; Depression | interventions — tianeptine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): Tianeptine
  Interventions: Drug: tianeptine

INTERVENTIONS:
Drug: tianeptine — tianeptine 12,5mg TID
  Other Names: Stablon (Servier)
  Arms: 2
Drug: Placebo — Placebo 12.5 mg TID
  Arms: 1

SUMMARY:
One of the main challenges in the treatment of Bipolar Disorder (BD) is to achieve better functioning outcomes after syndromal recovery. Even treatment-responsive patients, who remain symptomatically well for extended periods of time, frequently demonstrate sub-threshold symptoms and continuing psychosocial morbidity and cognitive impairment. The cognitive impairment that persists during interepisode periods stands out as a major correlate of functional impairment, and may be a core aspect of the BD pathophysiology.

In this context, tianeptine stands out as a therapeutic agent with unique properties, which match most of the conditions found in BD.

This is an enriched maintenance study of the use of tianeptine as an adjunctive therapy in bipolar depression. All participants will receive tianeptine in an open label manner for a period of two months, following which they will be assigned randomly to the treatment with tianeptine or placebo in a double-blind fashion for six months. All patients will remain on treatment as usual for the duration of the trial. Along with clinical response, the investigators will prospectively evaluate the improvement in working and declarative memory, two cognitive prefrontal- and hippocampus-dependent processes, respectively, and the effects of tianeptine on serum BDNF levels.

DETAILED DESCRIPTION:
One of the main challenges in the treatment of Bipolar Disorder (BD) is to achieve better functioning outcomes after syndromal recovery. Available treatments are reasonably effective in reducing acute symptoms, but many times the syndromal recovery is not accompanied by the restoration of functioning capabilities. This is particularly true for bipolar depression, which is responsible for most of the burden associated with BD. Even treatment-responsive patients, who remain symptomatically well for extended periods of time, frequently demonstrate sub-threshold symptoms and continuing psychosocial morbidity and cognitive impairment. The cognitive impairment that persists during interepisode periods stands out as a major correlate of functional impairment, and may be a core aspect of the BD pathophysiology. Beyond that, cognitive impairment worsens with cumulative episodes.

Functional and morphometric studies have shown changes in amygdala, hippocampus and prefrontal cortex of patients with bipolar disorder. Effective treatments for bipolar disorder, such as lithium and divalproex, have proved to prevent cellular atrophy, to have antiapoptotic properties and to increase BDNF levels. Findings from neuropathological studies have confirmed reduction and dysgenesis of neuronal cell lines in the hippocampus in bipolar disorder. Ultimately, a main challenge in the treatment of BD is translating the knowledge of neuronal plasticity and neurobiology of the illness into novel therapeutic options.

In this context, tianeptine stands out as a therapeutic agent with unique properties, which match most of the conditions found in BD. The neurochemical properties of tianeptine vary from those of other tricyclic and non-tricyclic antidepressants. Noteworthy, none of current available medications for BD showed all these features: 1) tianeptine exert opposite effects than chronic stress in neurons, increasing neuroprotective factors what may help to quench the cycle of affective episode recurrence and neural and deterioration; 2) tianeptine affects neuroplasticity in the hippocampus and have been reported to increase dendritic lengths; 3) tianeptine increases BDNF levels in the amygdala; 4) tianeptine attenuated stress-induced glutamate release in amygdala; 5) tianeptine has anticonvulsant properties via adenosinergic A1 receptors; 6) tianeptine has analgesic effects.

In the present research project, we plan on conducting an enriched maintenance study of the use of tianeptine as an adjunctive therapy in bipolar depression. All participants will receive tianeptine in an open label manner for a period of two months, following which they will be assigned randomly to the treatment with tianeptine or placebo in a double-blind fashion for six months. All patients will remain on treatment as usual for the duration of the trial. This trial will allow the investigation of the efficacy and tolerability of tianeptine 37.5mg/day as an adjunctive treatment of bipolar depression and its impact on clinical variables associated with the aftermath of a bipolar depression episode. Considering that tianeptine is approved to be used orally in humans and has been on the market for depression, a low risk intervention using a novel approach may be provided by this clinical trial. Along with clinical response, we will prospectively evaluate the improvement in working and declarative memory, two cognitive prefrontal- and hippocampus-dependent processes, respectively, and the effects of tianeptine on serum BDNF levels.

ELIGIBILITY:
Inclusion Criteria:

* To be included patients will be required to:

  * Meet DSM-IV criteria for bipolar disorder types I or II
  * Have current symptoms of depression, with a MADRS score over 12 at baseline
  * Have the capacity to consent to the study and comply with the study procedures
  * Use effective contraception in the case of women of childbearing age
  * Patients will need to be in a stable dose of mood stabilizer for at least one month prior to randomization.

Exclusion Criteria:

* Exclusion from the trial includes:

  * Patients with a well defined or suspected clinically unstable systemic medical conditions
  * Pregnant or lactating women
  * Patients who are currently taking augmentation medications or supplementation
  * Patients who do not tolerate the use of tianeptine
  * Inability to comply with either the requirements or informed consent of the treatment protocol.
* Withdrawal criteria:
* Withdrawal from the trial will take place whenever:

  * Patients stop taking medication or are deemed as non compliant by the attending physician
  * Patients stop taking contraceptives of become pregnant
  * Dose changes or additions/exclusions to existing medication - patients will be kept in the trial, but such changes will be computed as a primary outcome
  * Serious adverse reactions
  * Withdrawal of consent by the patient
  * Hospitalization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in mood symptoms (Hamilton depression rating scale) | @ 4 weeks and @ 8 months

SECONDARY OUTCOMES:
Cognitive improvement | @ 4 weeks and @ 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Kapczinski, MD,PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre and UFRGS
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil